CLINICAL TRIAL: NCT06331429
Title: Smart Technology Platform for Socio-emotional Development and Health Promotion: Implementation and Validation of a Serious Game in Adolescentes With DM1
Brief Title: Emoticare: Serious Game for the Adaptation to the Disease of Adolescents With Type 1 Diabetes Mellitus.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Universitat Politècnica de València (Other)
Responsible Party: Principal Investigator, M. Antonia Pérez-Marín, Associate Professor, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EmoTiCare
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes; Adolescent Development
Keywords: Type 1 Diabetes; Serious Game; Technology platform; Psychological intervention; Adolescence; Quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Patients who receive the treatment program, will previously constitute their own control group (waiting list control group).
- Experimental group (Experimental): Adolescents who receive the treatment program, will previously constitute their own control group (waiting list control group). Thus, diagnostic measures will be obtained in all of them in an initial evaluation (T1), and after 6 weeks of this assessment the treatment program will be started. In the first contact session at 6 weeks after T1 all adolescents will be re-assessed (T2) and after this the treatment program will be started (within an estimated time of 15 days maximum from this second pre-treatment evaluation, the estimated duration of treatment being 6 weeks). After the completion of the serious game, a new asssesment pass will be performed (T3) in order to assess the post-treatment change. Thus, the estimated time between T2 and T3 will be equivalent to that between T1 and T2, being 6 weeks.
  Interventions: Behavioral: EmoTiCare

INTERVENTIONS:
Behavioral: EmoTiCare — The EMOTICARE technological platform intervenes in users through a serious game, i.e. a video game whose main purpose is to teach or provide the player with certain skills that serve to achieve a higher purpose than the game itself.
  The game works in 6 areas, each of which refers to one of the variables that are analysed or considered important in the adaptation to the disease: Area 1. Psychoeducation of DM1; 2. Emotional awareness and expression; 3. Emotional regulation; 4. Problem solving; 5. Self-esteem and identity;6. Social skills and communication
  Arms: Experimental group

SUMMARY:
The intervention program targets adolescents with chronic Type 1 Diabetes Mellitus. Given the critical developmental stage and life transitions, necessitating robust personal resources, psychological support becomes imperative. To foster socioemotional skills and overall well-being, particularly crucial for averting future emotional issues and promoting a healthier, more fulfilling life, this support is especially vital for those dealing with chronic illnesses. Such conditions pose a risk for psychological problems, potentially complicating treatment and prognosis. Presently, digital and technological platforms are integrating psychological interventions for patients with chronic diseases, showcasing an innovative approach to address psychological challenges.

The platform integrates new technologies for assessment and intervention. Ecological Momentary Assessment enables real-time evaluation, with data transferred to the technological platform. Artificial intelligence personalizes interventions based on participants' socio-demographic characteristics and assessment results. Ecological Momentary Intervention is employed for in-context treatments in participants' daily lives and natural environments. A serious game method, proven effective in various interventions, is used to engage adolescents and young people intrinsically. The game encompasses six main areas aligning with theoretical models, facilitating the development of socio-emotional competencies, and promoting physical and psychological health. It addresses different aspects of psychological and subjective well-being, reinforcing resources needed to navigate vital changes in these developmental stages, especially when living with a chronic illness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Diabetes mellitus type 1 (6 months from diagnosis)
* Informed consent by parents/guardians and participants

Exclusion Criteria:

* Diagnosis other than type 1 diabetes mellitus
* No access to internet or new technologies
* Not speaking Spanish

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change Quality of Life (Baseline-Pre-Post) | Baseline up to 12 weeks
  KIDSCREEN-27. This scale consists of 27 items in 5 subscales. Physical well-being, mood, family life, school life, peer relations. Scores range from 27 to 135. Higher scores indicate a higher quality of life in general and in each of the subscales.
  First measurement: After the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 weeks after the first measurement, the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 weeks after the second measurement, the third measurement of the same variable was carried out.
Change Emotional and Behavioral Problems (Baseline-Pre-Post) | Baseline up to 12 weeks
  SDQ: This questionnaire is used to assess the possible presence of psychopathology and the emotional and behavioural adjustment of adolescents. It is a 25-item Likert-type (1-3) questionnaire. The items of this questionnaire are divided into 5 subscales: emotional symptomatology, conduct problems, hyperactivity, peer problems and prosocial behaviour. Higher scores on each scale indicate greater difficulties. First measurement: After the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 weeks after the first measurement, the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 weeks after the second measurement, the third measurement of the same variable was carried out.
Change Emotional Competences (Baseline-Pre-Post) | Baseline up to 12 weeks
  EAQ-30: This questionnaire consists of 30 Likert-style items (1-False to 3-True), and aims to identify how adolescents think about their feelings, as well as the degree to which they feel them and the ability to express them. In addition to an overall score, this tool is composed of 6 subscales that attempt to describe different aspects of emotional functioning. Higher scores indicate greater use of emotional awareness and regulation strategies.
  First measurement: After the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 weeks after the first measurement, the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 weeks after the second measurement, the third measurement of the same variable was carried out.
Change Self-concept (Baseline-Pre-Post) | Baseline up to 12 weeks
  CAG: This questionnaire aims to measure self-concept in adolescents from a multidimensional perspective. It consists of 48 Likert-type response items ranging from 1 to 5, providing a score range of 48 to 240. Physical Self-Concept, Social Acceptance, Family Self-Concept, Intellectual Self-Concept, Personal Self-Assessment, and Sense of Control. The questionnaire provides an overall self-concept score, as well as scores for 6 subdimensions: Higher scores indicate higher self-concept.
  This is the first measurement. After obtaining the participant's informed consent, we assessed the initial score for this outcome.
  The second measurement, labeled PRE, was conducted up to 6 weeks after the first measurement of the same variable.
  The third measurement, labeled POST, was carried out up to 6 weeks after the second measurement.
Change Coping (Baseline-Pre-Post) | Baseline up to 12 weeks
  Social Problem Solving Inventory- Revised (SPSI-R). This questionnaire attempts to reflect the cognitive, affective and behavioural responses to the problems of daily life or the different difficulties we try to solve. This reduced version consists of 25 Likert-type items, grouped into the following 5 dimensions: Rational problem solving, Avoidant style, Impulsive style, Positive problem orientation and Negative problem orientation. Higher scores on each dimension signify the coping style used by the adolescent.
  First measurement: After the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 weeks after the first measurement, the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 weeks after the second measurement, the third measurement of the same variable was carried out.
Change Social Skills (Baseline-Pre-Post) | Baseline up to 12 weeks
  CHASO: It consists of 40 Likert-type response items ranging from 1 to 5 (1 - Very uncharacteristic of me; 5 - Very characteristic of me) and assesses a total of 10 skills: 1. Interacting with strangers; 2. Dealing with criticism; 4. Interacting with people I am attracted to; 5. Staying calm in the face of criticism; 6. Public speaking/interacting with superiors; 7. The scores for each of these skills are calculated from the sum of the items that make them up. Higher scores indicate higher social skills.
  First measurement: After the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 weeks after the first measurement, the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 weeks after the second measurement, the third measurement of the same variable was carried out.

SECONDARY OUTCOMES:
Change Threat of disease(Baseline-Pre-Post) | Baseline up to 12 weeks
  The Brief Illness Threat Questionnaire (BIP-Q) is used, which consists of 5 items with a Likert scale from 0 to 10. This questionnaire mainly assesses consequences of the illness, duration of the illness, identity, worry about the illness and emotional impact of the illness. The scale is interpreted so that the higher the score, the greater the sense of perceived threat.
  First measurement: After the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 weeks after the first measurement, the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 weeks after the second measurement, the third measurement of the same variable was carried out.
Change Psychoeducation Diabetes | Start of the game and during the game
  Psychoeducation of the disease: the ECODI Diabetes knowledge scale will be used to assess this variable. This scale consists of 25 items and four dimensions: basic knowledge and self-care, laboratory values, diet and physical exercise. It is a scale that is corrected by the number of hits and misses.
  Psychoeducation about the disease: The ECODI diabetes knowledge scale is used to assess this variable. This scale consists of 25 items and four dimensions: basic knowledge and self-care, laboratory values, diet and exercise. It is a scale that is corrected by the number of hits and misses.
Change Resilience (Baseline-Pre-Post) | Baseline up to 12 weeks
  Connor-Davidson Resilience Scale to assess the ability to cope with stress and adversity. The resilience scale is made up of 10 items, with a range of scores from 0 to 40, with higher scores indicating greater resilience.
  First measurement: Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: PRE- Up to 6 weeks after the first measurement the second measurement of the same variable was carried out.
  Third measurement: POST Up to 6 weeks after the second measurement the third measurement of the same variable was carried out.

OTHER OUTCOMES:
Glycaemic control (Baseline-Pre-Post) | Baseline up to 12 weeks
  HbA1c: It will be used to evaluate the glycemic control of the diabetic patient in endocrinology diseases

CONTACTS AND LOCATIONS:
Overall Officials: Marián Pérez-Marín, PhD, Principal Investigator — University of Valencia
Locations (1):
- Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin-Avila J, Rodriguez-Jimenez E, Valero-Moreno S, Gil-Gomez JA, Montoya-Castilla I, Perez-Marin M. The impact of the emoTICare program on socioemotional adjustment and psychological well-being in adolescents with type 1 diabetes mellitus. Front Endocrinol (Lausanne). 2025 Oct 3;16:1668398. doi: 10.3389/fendo.2025.1668398. eCollection 2025. PMID 41113700